CLINICAL TRIAL: NCT04610905
Title: The Effect of Reducing Sedentary Behaviour in Comparison to Promoting Physical Activity on Chronic Non-specific Low Back Pain in a Sedentary Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment hampered
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Malfliet Anneleen, Assistant professor and postdoctoral researcher, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1432020000219
Record Dates: First submitted 2020-10-15; First posted 2020-11-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Chronic Low-back Pain; Sedentary Behavior
Keywords: sedentary behaviour; sedentary lifestyle; desk-bound; chronic pain; long-lasting pain
MeSH Terms: conditions — Sedentary Behavior; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): This group will be asked to maintain their daily routine.
- Reducing sedentary behavior (Experimental): This group needs to download an app on their computer and their smartphone. This app will give a notification every 30 minutes to walk during 2 minutes during working hours.
  Interventions: Behavioral: Reducing sedentary behaviour
- Increase physical activity (Experimental): This group will be asked to be more physically active. They need to be active during 150min/week. Additionnaly they need to be active in periods of at least 10 minutes.
  Interventions: Behavioral: Increase physical activity

INTERVENTIONS:
Behavioral: Reducing sedentary behaviour — This group needs to download an app on their computer and their smartphone. This app will give a notification every 30 minutes to walk during 2 minutes during working hours. The participants will receive a diary to write down whether they stand up.
  Arms: Reducing sedentary behavior
Behavioral: Increase physical activity — This group will be asked to be more physically active. They need to be active during 150min/week. It can include walking, to ride a bike, jogging, tennis, football,... Additionnaly they need to be active in periods of at least 10 minutes. The participants will receive a diary to write down which activity they did and also for how long.
  Arms: Increase physical activity

SUMMARY:
The investigators will recruit participants between the age of 18 and 65 with chronic non-specific low back pain and a sedentary lifestyle. The participants will be randomly assigned to one of the three groups. The first group is the control group, the participants will be asked to continue their daily routine. The second group is an intervention group, sedentary behaviour will be reduced. In the third group participants will be asked to increase their physical activity up to 150min/week. The intervention takes place over a period of 6 weeks. After the intervention the pressure pain threshold will be measured, average steps will be measured (accelerometer) and a questionnaire needs to be filled out. These results will be compared to the results before the intervention and to the results of the other groups.

DETAILED DESCRIPTION:
The investigators will recruit participants between the age of 18 and 65 with chronic non-specific low back pain and a sedentary lifestyle. The partcipants will be randomly assigned to one of the three groups. The first group is the control group, the participants will be asked to not change their daily routine. In the first intervention group sedentary behaviour will be reduced. The participants will be asked to download an app on their smartphone and computer. This app will ask the participants to stand up and walk during 2 minutes to interrupt their sedentary behaviour during working hours. In the second intervention group participants will be asked to increase their physical activity. More specifically the participants will be asked to be active for a period of 150min/week. The intervention takes place over a period of 6 weeks. During these 6 weeks the participants needs to wear an accelerometer the first and the last week of the intervention. The week before the intervention a pre-measurement will take place, this means that the participant needs to wear an accelerometer during a week, fill out a questionnaire (BPI and SF-36) and the pressure pain threshold will be measured. After the intervention (6 weeks) the pressure pain threshold will be measured, average steps will be measured (accelerometer) and a questionnaire needs to be filled out. These results will be compared to the results before the intervention and to the results of the other groups. With this study the investigators will investigate whether less sedentary behavior or more physical activity are beneficial for chronic low-back pain.

ELIGIBILITY:
Inclusion Criteria:

* CNLBP, for at least 3days/week for at least 3 months since the first symptoms.
* Failed back surgery syndrome is allowed (ie, more than 3 years ago, anatomically successful operation without symptom disappearance)
* Desk job, sedentary lifestyle (i.e. sitting for more than 6 hours per day). Given the greater risk of developing serious health problems when sitting for more than six hours a day.
* 18-65 years old
* Native Dutch speaker
* Refraining from analgesics, caffeine, alcohol or nicotine in the previous 48h of the assessments
* Not undertaking exercise (>3 metabolic equivalents) 3 days before the assessments
* Both sexes
* Experiencing chronic neck pain is allowed if CNLBP is the dominant complaint.

Exclusion Criteria:

* Any specific cause that can explain the CNLBP
* Physically demanding job (e.g. nurses, paramedics, construction workers,...)
* Chronic widespread pain (i.e. fibromyalgia, chronic fatigue syndrome)
* Chronic systematic diseases such as rheumatoid arthritis, diabetes, etc.
* Neuropathic pain
* Being pregnant or pregnancy (including giving birth) in the preceding year
* History of specific spinal surgery
* Cinical depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The Brief Pain Inventory (short form) | Baseline assessment (T0)
  Since chronic pain is a rather fluctuating condition, the question "Please rate your pain by circling the one number that best describes your pain on AVERAGE" is used as primary outcome measure to evaluate pain intensity. The answer to this question is formulated on an 11-point (i.e. 0-10) numeric rating scale (NRS), which is recommended as a core outcome measure in clinical trials of chronic pain. 0 indicates no pain, 10 indicates the worst pain imaginable.
The Brief Pain Inventory (short form) | Directly post-intervention (6 weeks after baseline assessement)
  Since chronic pain is a rather fluctuating condition, the question "Please rate your pain by circling the one number that best describes your pain on AVERAGE" is used as primary outcome measure to evaluate pain intensity. The answer to this question is formulated on an 11-point (i.e. 0-10) numeric rating scale (NRS), which is recommended as a core outcome measure in clinical trials of chronic pain. 0 indicates no pain, 10 indicates the worst pain imaginable.
The Brief Pain Inventory (short form) | 3 month follow-up
  Since chronic pain is a rather fluctuating condition, the question "Please rate your pain by circling the one number that best describes your pain on AVERAGE" is used as primary outcome measure to evaluate pain intensity. The answer to this question is formulated on an 11-point (i.e. 0-10) numeric rating scale (NRS), which is recommended as a core outcome measure in clinical trials of chronic pain. 0 indicates no pain, 10 indicates the worst pain imaginable.
The Brief Pain Inventory (short form) | 6 month follow-up (go/ no go principe = if there is still a difference in behaviour between the groups after 3 months, we organize a 6m follow-up)
  Since chronic pain is a rather fluctuating condition, the question "Please rate your pain by circling the one number that best describes your pain on AVERAGE" is used as primary outcome measure to evaluate pain intensity. The answer to this question is formulated on an 11-point (i.e. 0-10) numeric rating scale (NRS), which is recommended as a core outcome measure in clinical trials of chronic pain. 0 indicates no pain, 10 indicates the worst pain imaginable.

SECONDARY OUTCOMES:
Algometry (pressure pain threshold) | Baseline assessment (T0)
  Pressure pain thresholds will be assessed by using a handheld digital algometer. It evaluates the lowest stimulus in which a person perceives pain.
Algometry (pressure pain threshold) | Directly post-intervention (6 weeks after baseline assessement)
  Pressure pain thresholds will be assessed by using a handheld digital algometer. It evaluates the lowest stimulus in which a person perceives pain.
Algometry (pressure pain threshold) | 3 month follow-up
  Pressure pain thresholds will be assessed by using a handheld digital algometer. It evaluates the lowest stimulus in which a person perceives pain.
Algometry (pressure pain threshold) | 6 month follow-up. (go/ no go principe = if there is still a difference in behaviour between the groups after 3 months, we organize a 6m follow-up)
  Pressure pain thresholds will be assessed by using a handheld digital algometer. It evaluates the lowest stimulus in which a person perceives pain.
The Brief Pain Inventory (Short form) | Baseline Assessment (T0)
  The BPI is a questionnaire to assess pain severity and degree of interference in daily functioning. Scores range from 0 to 10, with higher scores indicating more pain, or more pain interference.
The Brief Pain Inventory (Short form) | Directly post-intervention (6 weeks after baseline assessement)
  The BPI is a questionnaire to assess pain severity and degree of interference in daily functioning. Scores range from 0 to 10, with higher scores indicating more pain, or more pain interference.
The Brief Pain Inventory (Short form) | 3 month follow-up
  The BPI is a questionnaire to assess pain severity and degree of interference in daily functioning. Scores range from 0 to 10, with higher scores indicating more pain, or more pain interference.
The Brief Pain Inventory (Short form) | 6 month follow-up (go/ no go principe = if there is still a difference in behaviour between the groups after 3 months, we organize a 6m follow-up)
  The BPI is a questionnaire to assess pain severity and degree of interference in daily functioning. Scores range from 0 to 10, with higher scores indicating more pain, or more pain interference.
Accelerometry (objective measures of physical activity and sedentary behavior) | Baseline assessment (T0)
  With a hip-worn accelerometer sedentary behavior and physical acitvity will be objectively measured.
Accelerometry (objective measures of physical activity and sedentary behavior) | Directly post-intervention (6 weeks after baseline assessement)
  With a hip-worn accelerometer sedentary behavior and physical acitvity will be objectively measured.
Short Form 36 Health Status Survey (SF-36) | Baseline assessment (T0)
  The SF-36 is a questionnaire to consider the health- related quality of life. Scores on the SF36 range from 0 to 400, with higher scores indicating better health.
Short Form 36 Health Status Survey (SF-36) | Directly post-intervention (6 weeks after baseline assessement)
  The SF-36 is a questionnaire to consider the health- related quality of life. Scores on the SF36 range from 0 to 400, with higher scores indicating better health.
Short Form 36 Health Status Survey (SF-36) | 3 month follow-up
  The SF-36 is a questionnaire to consider the health- related quality of life. Scores on the SF36 range from 0 to 400, with higher scores indicating better health.
Short Form 36 Health Status Survey (SF-36) | 6 month follow-up ( (go/ no go principe = if there is still a difference in behaviour between the groups after 3 months, we organize a 6m follow-up)
  The SF-36 is a questionnaire to consider the health- related quality of life. Scores on the SF36 range from 0 to 400, with higher scores indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: Anneleen Malfliet, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No